CLINICAL TRIAL: NCT05212896
Title: An Exploratory Clinical Study to Evaluate the Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of BC006 Monoclonal Antibody Injection in Patients With Advanced Solid Tumors Including Giant Cell Tumor of Tendon Sheath
Brief Title: An Exploratory Clinical Study of BC006 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dragonboat Biopharmaceutical Company Limited (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC006-Ⅰ-01
Record Dates: First submitted 2022-01-04; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-06

CONDITIONS: Advanced Solid Tumors (Including GCTTS)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: Phase Ia (Experimental): Participants will receive escalating doses of BC006 at assigned dose (0.08, 0.3, 1.0, 3.0, 10, 20 mg/kg) via intravenous (IV) infusion every 2 weeks until disease progression, unacceptable toxicity, withdrawal of informed consent, or up to 48 weeks of treatment, whichever occurs first.
  Interventions: Drug: BC006
- Dose Expansion: Phase Ib Cohort 1 (Experimental): Participants with GCTTS will receive BC006 at recommended dose for expansion (RDE) IV every 2 weeks until disease progression, unacceptable toxicity, withdrawal of informed consent, or up to 24 weeks of treatment, whichever occurs first.
  Interventions: Drug: BC006
- Dose Expansion: Phase Ib Cohort 2~4 (Experimental): Participants with other solid tumors will receive BC006 at RDE IV every 2 weeks until disease progression, unacceptable toxicity, withdrawal of informed consent, or up to 48 weeks of treatment, whichever occurs first.
  Interventions: Drug: BC006

INTERVENTIONS:
Drug: BC006 — BC006 monoclonal antibody injection

SUMMARY:
This is a first in human, open-label, exploratory phase I clinical study including dose escalation (Ia) and dose expansion (Ib) stage. It aims to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of BC006 in giant cell tumor of tendon sheath (GCTTS) and other advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent form.
2. Age ≥ 18 years.
3. Clinical diagnosis:

   Dose Escalation: Phase Ia
   * Histologically or cytologically confirmed GCTTS: initial treatment unresectable, or postoperative recurrence unresectable, or refuse surgical treatment.
   * Patients with histologically or cytologically confirmed advanced solid tumor, who have progression after prior SOC therapy, or who intolerant to SOC, or for whom there is no SOC therapy available.

   Dose Expansion: Phase Ib
   * Cohort 1: Histologically or cytologically confirmed GCTTS: initial treatment unresectable, or postoperative recurrence unresectable, or refuse surgical treatment.
   * Cohort 2~4: Patients with histologically or cytologically confirmed advanced solid tumor which is sensitive to Ia treatment，who have progression after prior SOC therapy, or who intolerant to SOC, or for whom there is no SOC therapy available.
4. Life expectancy ≥ 12 weeks.
5. Ia: at least one evaluable lesion; Ib: at least one measureable lesion as defined by RECIST V1.1.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
7. Evidence of adequate organ function by standard laboratory tests:

   * Adequate hematological function: Hemoglobin (Hgb) ≥ 90 g/L, Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, Platelets (Plts) ≥ 90 × 109/L.
   * Adequate liver function: Total bilirubin ≤ 1.5 × the upper limit of normal (ULN), Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) ≤ 2.5 × ULN (AST≤ 5 × ULN, ALT≤ 5 × ULN for subjects with liver metastases).
   * Adequate renal function: Creatinine ≤ 1.5 × ULN, or Creatinine clearance by Cockcroft Gault formula ≥ 50 mL/min.
   * Adequate Coagulation function: Activated partial thrombin time (APTT) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN, international standardized ratio (INR) ≤ 1.5 × ULN.
8. Female patients of child-bearing potential or male patients with a female partner(s) of child-bearing potential must agree to use reliable contraceptive methods (hormonal, condoms or abstinence) for the duration of the study and for 6 months after the last dose of BC006; women of child-bearing potential must have a negative blood or urine pregnancy test within 7 days prior to enrollment.

Key Exclusion Criteria:

1. Prior anti-tumor therapies such as radiotherapy, chemotherapy, targeted therapy, endocrine therapy, immunotherapy or other investigational agents within 4 weeks before the first dose of BC006.
2. Prior treatment with any anti-CSF-1R inhibitor.
3. Any toxicity from previous anti-tumor treatments have not recovered to CTCAE V5.0 grade ≤ 1 (except treatment-related alopecia).
4. Patients with untreated or clinically symptomatic brain metastases, spinal cord compression, cancerous meningitis, or patients with evidence that brain and spinal cord metastases have not been controlled (Patients with previously treated brain metastases may participate provided they are clinically and imaging stable for at least 4 weeks prior to first dose of BC006, have no evidence of cerebral edema and are off steroids).
5. Patients with severe cardiovascular diseases: cardiac arrhythmia requiring clinical intervention; acute coronary syndrome, congestive heart failure, stroke or other ≥ grade 3 cardiovascular events within 6 months; New York Heart Association (NYHA) cardiac function ≥ grade II or left ventricular ejection fraction (LVEF) <50%; poorly controlled hypertension as judged by the investigator are not suitable to participate in the study.
6. Receipt of a live vaccine within 4 weeks prior to the first dose of BC006 or anticipation that such a live vaccine will be required during the study.
7. Patients with symptomatic pleural, abdominal, or pericardial effusions that require repeated puncture and drainage treatment and cannot be relieved; patients with stable disease after receiving treatment (including therapeutic thoracentesis or abdominal puncture) are allowed to enroll.
8. In the opinion of the investigator, patients have any clinical or laboratory examination abnormality or other conditions that are not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-limiting Toxicities (DLTs) | Up to 28 days
  Dose Escalation: Phase Ia
Maximum Tolerated Dose (MTD) of BC006 | Up to 28 days
  Dose Escalation: Phase Ia
Recommended Dose for Expansion (RDE) of BC006 | Through study completion, an average of 1 year
  Dose Escalation: Phase Ia
Number of Participants with TEAEs | Through study completion, an average of 1 year
  Graded according to the NCI CTCAE V5.0
Number of Participants with SAEs | Through study completion, an average of 1 year
  Graded according to the NCI CTCAE V5.0

SECONDARY OUTCOMES:
Cmax | From first dose of BC006, an average of 6 months
  Pharmacokinetic parameter, observed Maximum Serum Concentration (Cmax) of BC006
Tmax | From first dose of BC006, an average of 6 months
  Pharmacokinetic parameter, Time-to-Maximum (Tmax) of BC006
AUC0-t | From first dose of BC006, an average of 6 months
  Pharmacokinetic parameter, area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration (AUC0-t) of BC006
t1/2 | From first dose of BC006, an average of 6 months
  Pharmacokinetic parameters, apparent Terminal Half-life (t1/2) of BC006
Pharmacodynamic (PD) Parameters | From first dose of BC006, an average of 6 months
  CSF-1 levels in peripheral blood
Number of Participants with Anti-BC006 Antibodies (ADAs) | From first dose of BC006, an average of 6 months
  ADA titer and Neutralizing Antibodies (NAbs) analysis will be performed when ADA is positive
Objective Response Rate (ORR) | From first dose of BC006, up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Disease Control Rate (DCR) | From first dose of BC006, up to 2 years
  Disease control rate (DCR) is defined as the proportion of the optimal time response of CR, PR, disease stable (SD) (i.e. CR+PR+SD) between initiation of the trial drug and withdrawal from the trial, as assessed according to RECIST Version 1.1
Progression-Free Survival (PFS) | From first dose of BC006, up to 2 years
  Progression-free survival (PFS) is defined as the time elapsed from the day the study drug was first administered until the first imaging assessment of disease progression (PD) or death from any cause.
Duration of Response (DOR) | From first dose of BC006, up to 2 years
  The duration of response (DOR) is defined as the time from the beginning of the first tumor assessment as PR or CR to the first assessment as PD or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zheng, Study Chair — West China Hospital
Locations (1):
- Dragonboat Biopharmaceutical,Co.,Ltd, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No